CLINICAL TRIAL: NCT02939430
Title: Sugammadex Reversal of Neuromuscular Blockade and Postoperative Bleeding
Acronym: Suga_bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, lecturer of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Refa-suga-bleeding
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Blood Coagulation Tests ( INR, APTT)
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Reversal of neuromuscular blockade will be performed using classic drugs (neostigmine 80 mic/kg and atropine 40 mic/kg)
  Interventions: Drug: Intravenous neostigmine and atropine
- Sugammadex group (Experimental): Reversal of neuromuscular blockade will be performed using Sugammadex 2mg/kg
  Interventions: Drug: Sugammadex intravenous

INTERVENTIONS:
Drug: Sugammadex intravenous — Intravenous Injection of sugammadex (2 mg/kg) for reversal of rocuronium induced muscle relaxation
  Arms: Sugammadex group
Drug: Intravenous neostigmine and atropine
  Arms: Control

SUMMARY:
Sugammadex is new drug that is used for reversal of rocuronium induced muscle relaxation. benefits of reversal of neuromuscular blockade appears to be of great value in living donor liver transplant recipients. However, Few Clinical reports have investigated the anticoagulant effect of sugammadex. In this study, effects of sugammadex on bleeding profile of living donor liver transplantation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* all candidates for living donor liver transplantation

Exclusion Criteria:

* massive intraoperative bleeding manifestations of early graft dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
activated partial thromboplastin tile in seconds | 30 min

SECONDARY OUTCOMES:
international normalized ratio in second | 30 min

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university, Al Mansurah, Dkahleya
  - Gastroenterology center, Al Mansurah

IPD SHARING:
Plan to Share IPD: Yes